CLINICAL TRIAL: NCT06389604
Title: Preparing for Heat Waves - Enhancing Human Thermophysiological Resilience
Acronym: Prep4heat
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NL86367.068.24
Record Dates: First submitted 2024-03-05; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Body Temperature Changes; Heat Exposure; Heat Stress; Hyperthermia
Keywords: heat acclimation; thermoregulation; heat exposure; cardiovascular
MeSH Terms: conditions — Body Temperature Changes; Heat Stress Disorders; Hyperthermia

STUDY DESIGN:
Intervention Model Description: Non-randomized, within subject experiemental trial
Masking Description: No blinding due to nature of intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heat acclimation (Experimental): Passive heat exposure (29-35ºC; 6h/day for 7 days) in combination with 30min/day low-to-moderate intensity cycling.
  Interventions: Other: Heat acclimation

INTERVENTIONS:
Other: Heat acclimation — Daily repeated heat exposure to assess the effects of combined passive and active heat acclimation

SUMMARY:
As the ongoing progression of climate change exposes individuals to elevated temperatures and an escalating frequency of extreme heat events, the risk of more intense and prolonged heat waves raises significant concerns for public health, particularly among vulnerable populations. The physiological response to acute heat stress involves involuntary thermolytic reactions that may strain the cardiovascular system, especially in individuals with pre-existing vulnerabilities. Heat acclimation has been identified as a potential strategy to enhance thermoregulation and mitigate the adverse effects of heat stress. While existing research primarily focuses on athletes and military, this study aims to investigate the impact of a practical heat acclimation strategy, combining passive and active heat exposure, on thermophysiological, cardiovascular and metabolic parameters in healthy overweight adults. The study targets a population at increased risk for heat-related complications, seeking to provide realistic guidelines for broader application when a heat wave appears on the weather forecast.

DETAILED DESCRIPTION:
A non-randomized, within-subject experimental trial will be conducted. The complete study will consist of a screening day, a control week, a heat acclimation week, 3 heat stress test (HST) and meal-test (MT) days (t = -7, 0, and 8 (days)). To avoid a confounding effect of seasonal thermal differences and achieve maximal methodological quality, the study will be performed in the shortest possible timeframe for each participant. Given the seasonal fluctuations in NL, transitioning from April (~7oC) to June (~20oC), a crossover design is not applicable as a washout period of approximately 2 months would be needed and the measurements would likely take place in different climatic outdoor conditions. In total, 12 healthy male and female participants will be included in the study. During the no-intervention week (week 1), participants will be asked to continue their normal life at home, without being present at the university. In addition, during week 1, participants will be asked to wear a temperature sensor on their clothing to measure the environment temperature they are exposed to at home. Thereafter, on the intervention week (week 2), participants will be exposed to increasing elevated temperatures and undergo 30 min of low-to-moderate intensity cycling in the heated laboratory room for 7 days. The temperature settings are derived from past heat waves in the Netherlands, ensuring a realistic representation. The low exercise intensity is selected to be accessible to the majority of individuals within the target population. The HST-MT will be conducted on the first visit after the screening to serve as baseline measurements. The same tests will also be repeated before and after the heat acclimation week to determine the physiological response to increasing ambient temperatures. All measurements will take place in the Metabolic Research Unit of Maastricht University (MRUM), the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* 60 to 80 years
* BMI 25-30 kg/m2
* Sedentary (<2h exercise/week)

Exclusion Criteria:

* Presence of chronic cardiovascular disease, as determined by medical history and physical examination
* Participating in a structured exercise program
* Taking hot baths/saunas regularly
* Travelled for a prolonged time to destinations with elevated temperatures the last 3 months
* Pre-existing T2DM
* Blood donation within a month of study initiation
* People with low haemoglobin concentration (males: Hb = 13.5-17.5 g/dL, females: Hb = 11.5-15.5 g/dL)
* Recent participation in biomedical study (less than 1 month)
* Using any medication that may influence glucose or lipid metabolism (beta-blockers, thyroid medications, stimulants, antidepressants, anticoagulants)
* Smoking or abuse of alcohol

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Core temperature | 1 week of heat acclimation
  thermophysiological parameters (ºC)

SECONDARY OUTCOMES:
Skin temperature | 1 week of heat acclimation
  thermophysiological parameters (ºC)
Sweat rate | 1 week of heat acclimation
  thermophysiological parameters (mL/min)
Heart rate | 1 week of heat acclimation
  cardiovascular parameters (bpm)
Blood pressure | 1 week of heat acclimation
  cardiovascular parameters (mmHg)
Skin blood flow | 1 week of heat acclimation
  cardiovascular parameters (mL/min)
Energy expenditure | 1 week of heat acclimation
  Metabolic parameters (kJ/min)
Substrate oxidation | 1 week of heat acclimation
  glucose and fat oxidation (umol/kg/min)
Plasma metabolites | 1 week of heat acclimation
  Plasma glucose, insulin, free-fatty acids, triglycerides, total cholesterol (mmol/L)
Brain blood flow | 1 week of heat acclimation
  additional cardiovascular parameters (mL/min)
Flow-mediated dilation | 1 week of heat acclimation
  endothelial function, (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Pallubinsky, Dr., Principal Investigator — Maastricht University; Guy Plasqui, Principal Investigator — Maastricht University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pallubinsky H, Schellen L, Kingma BRM, Dautzenberg B, van Baak MA, van Marken Lichtenbelt WD. Thermophysiological adaptations to passive mild heat acclimation. Temperature (Austin). 2017 Mar 10;4(2):176-186. doi: 10.1080/23328940.2017.1303562. eCollection 2017. PMID 28680933
- [Background] Pallubinsky H, Phielix E, Dautzenberg B, Schaart G, Connell NJ, de Wit-Verheggen V, Havekes B, van Baak MA, Schrauwen P, van Marken Lichtenbelt WD. Passive exposure to heat improves glucose metabolism in overweight humans. Acta Physiol (Oxf). 2020 Aug;229(4):e13488. doi: 10.1111/apha.13488. Epub 2020 Jun 1. PMID 32359193